CLINICAL TRIAL: NCT05142878
Title: Pressure Ulcer Prevention Using Static Air Foam Hybrid Mattress (Ultracore Repose®) in a High Risk Population in Nursing Homes: A Multi-Center Cohort and Qualitative Study
Brief Title: What is the Incidence of Pressure Ulcer Category II-IV (Including Deep-tissue Injury and Unstageable) on a Static Air Foam Hybrid Mattress?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Frontier Medical Group, UK (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EC/2020/BC-06758; EC/2020/BC-06758 (Other: Ethics Committee UZ Ghent)
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Pressure Ulcer; Pressure Injury; Pressure Sore; Bed Sore
Keywords: static air support devices; High risk population; Elderly; Prevention; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Static air support devices (Ultracore Repose®) (Experimental): Residents will be placed on a static air foam hybrid mattress during 14 days:
  • Ultracore Repose® Mattress
  Interventions: Device: Ultracore Repose® mattress

INTERVENTIONS:
Device: Ultracore Repose® mattress — Residents will be placed on the Ultracore Repose® mattress during 14 days

SUMMARY:
Pressure ulcers are a serious and common problem for residents admitted to long-term care facilities and community care patients. They represent a major burden to patients, carers and the healthcare system, affecting approximately 1 in 20 community patients. They occur frequently among patients with limited mobility, such as those patients being bed-bound and/or wheelchair-bound. In many countries, pressure ulcers are recognized as a national health issue and governments designate pressure ulcers as one of the most important sentinel events for healthcare.

International guidelines recommend the use of pressure redistributing support surfaces, systematic patient repositioning and preventive skin care to prevent pressure ulcers. All interventions should be patient-tailored and based on a thorough assessment of both the patient and contextual risk factors. As pressure ulcers can arise in a number of ways, interventions for prevention and treatment need to be applied across a wide range of settings, including the community, nursing homes and hospitals.

A review of mortality and severe harm incidents reported to the National Reporting and Learning System found that pressure ulcers were the largest proportion of patient safety incidents in 2011/2012, accounting for 19% of all reports.

It has been acknowledged that a significant proportion of pressure ulcers are avoidable. The prevalence of pressure ulcers is 1 of the 4 common harms recorded in the UK NHS Safety Thermometer, a local improvement tool for measuring, monitoring and analysing patient harms across a range of settings, including nursing homes, community nursing and hospitals on a monthly basis.

Continuous low levels or short-term high levels of pressure and shear on the skin and underlying tissue on vulnerable areas are extrinsic factors contributing to the development of pressure ulcers. Support surfaces (e.g. any mattresses, integrated bed systems, mattress replacement, overlay, seat cushion, or seat cushion overlay) are specialized devices for pressure redistribution specifically designed for management of tissue loads, micro- climate, and/or therapeutic functions.

A Cochrane systematic review by McInnes et al. (2015) defined multiple groups of pressure redistribution materials: low-tech (not electrically driven) constant low-pressure supports, high-tech supported surfaces, and other supported surfaces (operating table mattress pad, rotating beds, cushions, and limb protectors). Static or reactive overlay mattresses are an example of a low-tech constant low pressure support. Static air mattresses maintain a continuous low air pressure that exerts a pressure redistributing effect. Serraes and Beeckman (2016) found a pressure ulcer incidence of 5.1% in patients placed on static air support surfaces (mattress overlay, heel wedge, and seat cushion) in a high risk population in a nursing home setting in Belgium.

A multicentre randomised controlled clinical trial in 26 nursing homes (including 308 residents) between April 2017 and May 2018 resulted in a significantly lower pressure ulcer incidence when applying the principle of static air (n=8/154, 5.2%) compared to the alternating air group (n=18/154, 11.7%)(p=0.04). The median time to develop a pressure ulcer category II-IV was significantly longer in the static air group (10.5 days, IQR 1-14) compared to the alternating air group (5.4 days, IQR 1-12; p=0.05). The study concluded that a static air mattress was significantly more effective compared to an alternating air pressure mattress to prevent pressure ulcers in a high risk nursing home population.

This multicentre cohort study will be performed in 5 nursing homes in a random sample of 40 residents who are at high risk of developing pressure ulcers. Residents will be included in the study for a period of 14 days. Skin assessment and risk factor registration will be done on a daily basis by the nurses. Reliability checks and time measurements will be completed by the researcher.

ELIGIBILITY:
Nursing home residents:

Inclusion criteria:

* High risk of pressure ulcers (Braden score < 12) and/or pressure ulcer category 1,
* Bedbound (> 8 hours in bed) or chair bound (> 8 hours in chair),
* Aged > 65 years,

Exclusion criteria:

* Pressure ulcer Category II-IV, deep tissue injury (DTI) or unstageable pressure ulcer,
* Expected length of stay < 2 weeks,
* End of life care,
* Medical contraindication for use of static air support devices

Caretakers:

Caretakers will be included in the focus group interviews if they have experience with the use of both the Ultracore Repose® mattress and the Repose overlay mattress®

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence (Cat. II+) | 14 days
  Incidence rate of pressure ulcers Cat. II-IV (including deep- tissue injury, unstageable), not associated with the use of medical devices

SECONDARY OUTCOMES:
Insight in caretakers' experiences and perceptions | 14 days
  Insight in caretakers' experiences and perceptions (outcome of the focus group interviews) after using Static Air Foam Hybrid Mattress

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Principal Investigator — University Ghent
Locations (5):
- Belgium (5):
  - WZC Egmont, Zottegem, Oost-Vlaanderen
  - WZC Heilig Hart, Oudenaarde, Osst-Vlaanderen
  - Woonzorgcentrum Ter Potterie, Bruges, West-Vlaanderen
  - Huize Zonnelied, Ieper, West-Vlaanderen
  - De Plataan, Izegem, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Website of the research group — http://www.ucvvgent.be